CLINICAL TRIAL: NCT01580215
Title: Long Term Follow up Investigation of Endobronchial Valves in Emphysema
Acronym: LIVE
Status: Terminated | Type: Observational
Why Stopped: Inability to reach desired recruitment goal; Sponsor executed other RCTs
Sponsor: Pulmonx International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Pulmonx Corporation (Industry)
Other Study IDs: 630-0013
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Pulmonary Emphysema
Keywords: Valves; Endobronchial; Endoscopic lung volume reduction; Pulmonx; Zephyr; Chartis; Emphysema; COPD
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Main cohort: * Patients of both genders of at least 18 years of age
  * Who understand and voluntarily sign an informed consent form
  * FEV1 > 15% predicted and < 45% predicted
  * RV >180% predicted
  * Diagnosis of emphysema with CT evidence of hyperinflation
  * Absence of collateral ventilation according to Chartis Assessment System
  * Treated with Zephyr Endobronchial Valve (EBV)
  Interventions: Device: Zephyr Endobronchial Valve (EBV)

INTERVENTIONS:
Device: Zephyr Endobronchial Valve (EBV) — • Implantation of at least one Zephyr EBV following Chartis assessment

SUMMARY:
This is an observational prospective single arm multicentre study to observe the effect over 5 years of Zephyr endobronchial valve therapy for emphysema.

DETAILED DESCRIPTION:
Primary objective is pulmonary function as assessed by FEV1 and secondary objectives are health related quality of life as assessed by the modified MRC dyspnea score and by the COPD assessment test, and survival at five years. 2000 patients will be enrolled in the study from approximately 200 referring centres in Germany. Patients will be followed up at 3, 6, and 12 months, and then yearly up to 5 years. The study will observe normal clinical practice. No investigations beyond those performed in normal clinical practice will be required with the exception of two short questionnaires. Patients will only be enrolled in the study if they have provided informed written consent for their anonymised data to be used in the study. Zephyr Endobronchial Valve has CE mark and is fully reimbursed in Germany and will not be provided by the sponsor for this study but will be obtained through normal commercial channels in accordance with normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders of at least 18 years of age
* Understand and voluntarily sign an informed consent form.
* FEV1 > 15% predicted and < 45% predicted
* RV >180% predicted
* Diagnosis of emphysema with CT evidence of hyperinflation . Absence of collateral ventilation according to Chartis Assessment System

Exclusion Criteria:

• Active pulmonary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient participation is entirely voluntary. Patients must meet the inclusion/exlusion criteria to be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2012-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
FEV1 | 2 years
  Relative (percentage) change from baseline at 2 years (24 months) of the Forced Expiratory Volume in one second (FEV1)

SECONDARY OUTCOMES:
Modified Medical Research Council (mMRC) Questionnaire | 5 years
  Absolute and relative change from baseline at each visit over the 5 year period of the Modified Medical Research Council (mMRC) Score
COPD Assessment Test (CAT) | 5 years
  Absolute and relative change from baseline at each visit over the 5-year period for the COPD Assessment Test (CAT)
Survival over 5 years | 5 years
  Survival status over the 5 year study period

OTHER OUTCOMES:
Adverse Events | 5 years
  Tabulation of adverse events occuring over the 5 year study period

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, Prof. Dr., Principal Investigator — Medizinische Fakultät Heidelberg
Locations (1):
- Heidelberg Hospital, Heidelberg, Germany